CLINICAL TRIAL: NCT00204542
Title: Comparison of the Efficacy and Tolerability of Solaraze for 3 vs. 6 Months in Patients With Mild to Moderate Actinic Keratosis Located at the Face and Head
Brief Title: Comparison of the Efficacy and Tolerability of Solaraze for 3 Versus 6 Months in Patients With Mild to Moderate Actinic Keratosis Located on the Face and Head
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Prof. Dr. Claus Garbe, DECOG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADO-Solaraze-AK-3-6; Eudra-CT-Nr. 2004-002761-21
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2009-03

CONDITIONS: Photosensitivity Disorders
Keywords: actinic keratosis; diclofenac sodium
MeSH Terms: conditions — Photosensitivity Disorders; Keratosis, Actinic | interventions — Diclofenac

ARMS (2):
- A (Active Comparator): Solaraze(R) 2x/day for 3 months
  Interventions: Drug: Diclofenac
- B (Active Comparator): Solaraze(R) 2x/day for 6 months
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac — Solaraze® (Diclofenac sodium) 2x/day topical for 3 months
  Arms: A
Drug: Diclofenac — Solaraze® (Diclofenac sodium) 2x/day topical for 6 months
  Arms: B

SUMMARY:
Topical treatment of mild to moderate actinic keratosis located on the face and head with Solaraze® is known to be a safe and efficient treatment option. However, it is unclear if an expansion of the treatment period to 6 months will increase the rate of complete responses.

Therefore the investigators will evaluate the efficacy and safety of the treatment of actinic keratosis with Solaraze® applied twice daily to the face and head over 3 or 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Visible and histologically proven actinic keratosis
* Prepared and able to give written informed consent
* ≥ 18 -80 years of age
* Prepared and comply with all study requirements, including the following: application of gel on the treatment area twice a day, 5 / 7 clinic visits during the prestudy, treatment, posttreatment, and follow-up period
* Pre- and posttreatment biopsy for histological confirmation (of clearance) of actinic keratosis diagnosis

Exclusion Criteria:

* Data of clinically significant, unstable, cardiovascular or haematologic, hepatic, neurologic, renal, endocrine, collagen-vascular, or gastrointestinal abnormalities or diseases
* Known allergies to any excipient in the study drug
* Any dermatological disease and/or condition in the treatment or surrounding area (3 cm distances from treatment area) that may be exacerbated by treatment with diclofenac or cause difficulty with examination
* Active chemical dependency or alcoholism, as assessed by the investigator
* Currently participating in another clinical study or have completed another clinical study with an investigational drug within the past 30 days
* Received topical treatment at the treatment area with imiquimod or 5-FU within a time period of 1 month
* Invasive tumours within the treatment area, e.g. merkel cell carcinoma, squamous cell carcinoma, basal cell carcinoma, the latter is accepted if completely surgically removed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2005-06; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Histologically controlled complete clearance of the actinic keratosis | 6 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, MD, Principal Investigator — Skin Cancer Program, Department of Dermatology, University Hospital Tübingen
Locations (4):
- Germany (4):
  - Skin Cancer Program, Department of Dermatology, Liebermeisterstrasse 8, Tübingen, Baden-Wurttemberg
  - Klinik fuer Dermatologie, Venerologie und Allergologie der Charite, Berlin
  - Dept. of Dermatology, Freiburg im Breisgau
  - Praxis Priv.-Doz. Dr. med. Dirschka, Wuppertal

REFERENCES:
- [Background] Nelson C, Rigel D, Smith S, Swanson N, Wolf J. Phase IV, open-label assessment of the treatment of actinic keratosis with 3.0% diclofenac sodium topical gel (Solaraze). J Drugs Dermatol. 2004 Jul-Aug;3(4):401-7. PMID 15303784
- [Background] Rivers JK. Topical 3% diclofenac in 2.5% hyaluronan gel for the treatment of actinic keratoses. Skin Therapy Lett. 2004 Jan;9(1):1-3. PMID 14716439
- See also: Link to published abstract — http://www.ncbi.nlm.nih.gov/pubmed/21414035